CLINICAL TRIAL: NCT06290349
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel, Phase III Clinical Trial to Evaluate the Efficacy and Safety of DA5221-T When Added to Ongoing DA5221-B1 and DA5221-B2 Combination Therapy in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control
Brief Title: Efficacy and Safety of DA5221-T When Added to Ongoing DA5221-B1 and DA5221-B2 Combination Therapy in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA5221_DM_III
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DA5221-T1 + DA5221-R2 + DA5221-B1 + DA5221-B2 (Experimental)
  Interventions: Drug: DA5221-T1; Drug: DA5221-B1; Drug: DA5221-B2
- DA5221-R1 + DA5221-T2 + DA5221-B1 + DA5221-B2 (Experimental)
  Interventions: Drug: DA5221-T2; Drug: DA5221-B1; Drug: DA5221-B2
- DA5221-R1 + DA5221-R2 + DA5221-B1 + DA5221-B2 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: DA5221-B1; Drug: DA5221-B2

INTERVENTIONS:
Drug: DA5221-T1 — DA5221-T1 + DA5221-R2, orally, once daily, up to 24 weeks
  Arms: DA5221-T1 + DA5221-R2 + DA5221-B1 + DA5221-B2
Drug: DA5221-T2 — DA5221-R1 + DA5221-T2, orally, once daily, up to 24 weeks
  Arms: DA5221-R1 + DA5221-T2 + DA5221-B1 + DA5221-B2
Drug: Placebo — DA5221-R1 + DA5221-R2, orally, once daily, up to 24 weeks
  Arms: DA5221-R1 + DA5221-R2 + DA5221-B1 + DA5221-B2
Drug: DA5221-B1 — DA5221-B1, orally, daily for background therapy
Drug: DA5221-B2 — DA5221-B2, orally, daily for background therapy

SUMMARY:
This study evaluates the efficacy and safety of adding the SGLT-2 inhibitor DA5221-T to the combination therapy of DA5221-B1 and the DPP-4 inhibitor DA5221-B2 in patients with type 2 diabetes who have inadequate blood glucose control. The study focuses on assessing the effectiveness and safety of the triple combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type II diabetes mellitus aged 19 years or older
2. Patients who had taken DA5221-B1 and DA5221-B2(or another DPP-4 inhibitor is allowed) combination therapy at the same dose for at least 8 weeks prior to the screening visit
3. Patients with fasting plasma glucose≤270mg/dL at the screening visit
4. Patients with 18.5kg/m^2≤BMI≤40kg/m^2 at the screening visit
5. Patients who have signed an informed consent themselves after receiving detailed explanation about the clinical study

Exclusion Criteria:

1. Patients with type 1 diabetes, secondary diabetes, gestational diabetes, diabetic coma or -pre-coma, metabolic acidosis including lactic acidosis and diabetic ketoacidosis
2. Patients with a medical history of New York Heart Association(NYHA) class III~IV heart failure or with congestive heart failure, acute and unstable heart failure
3. Patients with severe infectious disease or severe traumatic systemic disorders
4. Patients with hypopituitarism or adrenal insufficiency, pulmonary infarction, severe pulmonary dysfunction and other hypoxemia
5. Patients with galactose intolerance, lapp lactase deficiency, glucosegalactose malabsorption

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from the baseline in HbA1c (%) after 24 weeks | Baseline, 24 weeks

SECONDARY OUTCOMES:
Change from the baseline in fasting plasma glucose(mg/dL) after 24 weeks | Baseline, 24 weeks
Change from the baseline in HbA1c response rate(<7.0%, <6.5%) after 24 weeks | Baseline, 24 weeks
Change from the baseline in weight after 24 weeks | Baseline, 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University college of Medicine, Seoul, South Korea